CLINICAL TRIAL: NCT04717037
Title: Olive Oil Massage Effect for Reduction of Preterm Sepsis (OMEPS), Randomized Controlled Trial
Brief Title: Olive Oil Massage Effect for Reduction of Preterm Sepsis (OMEPS)
Acronym: OMEPS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: King Abdulaziz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RJ20/109/J
Record Dates: First submitted 2020-12-08; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Sepsis; Pre-Term; Late-Onset Neonatal Sepsis
Keywords: Olive oil; Massage; Preterm; Late-Onset sepsis
MeSH Terms: conditions — Sepsis; Premature Birth; Neonatal Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): The olive oil massage will be applied initially at 72 hrs of life then twice daily with a dose of 4ml/kg till 28 days .
  Interventions: Biological: Olive Oil Massage
- Control (No Intervention): Patients who are assigned to the control group will receive standard care as per unit policies.

INTERVENTIONS:
Biological: Olive Oil Massage — olive oil massage application.
  Arms: Study

SUMMARY:
The OMEPS trial is a randomized clinical trial in the western region of Saudi Arabia. Conducted to assess the safety and feasibility of olive oil as massage for preterm infants and if associated with reduced risk of Late-Onset sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants born at one of the participated centers.
2. Preterm Infants born at ≥24weeks gestation and ≤32weeks gestation
3. Birth weight ≥ 500gm up to 2000 gm.

Exclusion Criteria:

1. Outborn Infants.
2. Preterm infants < 24wk or > 32 wk
3. Preterm infants < 500 gm or > 2000gm
4. Critically ill patients, e.g., Hemodynamic unstable, culture-confirmed neonatal sepsis, Hydrops fetalis, Life-threatening congenital anomalies.
5. Congenital skin anomalies or infection
6. Major surgical procedure
7. Any patient whose parents refuse consent.
8. Death within 48 hours of life.

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of culture-proven sepsis in the blood or CSF | 72 hours from birth till 28 days of life
  Primary outcomes defined as the rate of culture-proven sepsis in the blood or CSF in the 28 days of life.Late-onset sepsis defined as sepsis onset after 72 h of life.
  The olive oil will be applied initially at 72 hours of life then twice daily with a dose of 4ml/kg.

SECONDARY OUTCOMES:
Neonatal Skin Condition score | 72 hours from birth till 28 days of life
  Validated Scoring system [ Neonatal Skin Condition Score ] will be used to score the skin integrity, and care will be monitored at baseline then weekly till age 28th of life or discharge.
  Skin condition was assessed with the Neonatal Skin Condition Score,This score has 9 scores from 1 to 9, 1 depicting the best skin state and 9 the worst with erythema, blistering & oozing over the entire area.

CONTACTS AND LOCATIONS:
Overall Officials: Jubara Alallah, Principal Investigator — King Abdulaziz Medical city , WR
Locations (2):
- Saudi Arabia (2):
  - King Abdulaziz Medical City, Jeddah, WR
  - King Abdulaziz University Hospital, Jeddah

IPD SHARING:
Plan to Share IPD: No